CLINICAL TRIAL: NCT01943305
Title: An Open-label Phase 2a Clinical Trial to Test the Effect of Yellow Fever Vaccination in a Background of Japanese Encephalitis Antibodies.
Brief Title: The Role of Pre-existing Cross-reactive Antibodies in Determining the Efficacy of Vaccination in Humans
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Singapore General Hospital (Other)
Collaborators: Duke-NUS Graduate Medical School (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: EID-JE/YF-01
Record Dates: First submitted 2013-09-03; First posted 2013-09-16 (Estimated); Last update posted 2016-04-20 (Estimated); Status verified 2016-04

CONDITIONS: Yellow Fever; Encephalitis, Japanese
Keywords: Yellow Fever; vaccination; Japanese encephalitis; antibodies
MeSH Terms: conditions — Yellow Fever; Encephalitis, Japanese | interventions — Japanese Encephalitis Vaccines; Yellow Fever Vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Test arm (Experimental): A total of 100 healthy adults, pre-screened to be negative for anti-dengue antibodies will be enrolled upon written informed consent. 75 subjects in the test arm will received 2 doses of inactivated Japanese Encephalitis vaccine and 1 dose of Yellow Fever vaccine.
  Interventions: Biological: Japanese Encephalitis vaccine; Biological: Yellow Fever vaccine
- Control arm (Experimental): A total of 100 healthy adults, pre-screened to be negative for anti-dengue antibodies will be enrolled upon written informed consent. 25 subjects in the control arm will not receive Japanese Encephalitis vaccine but will receive 1 dose of Yellow Fever vaccine.
  Interventions: Biological: Yellow Fever vaccine

INTERVENTIONS:
Biological: Japanese Encephalitis vaccine — IXIARO, inactivated, adsorbed vaccine. Two doses (0.5 ml each) of IXIARO one month apart
  Other Names: Ixiaro
  Arms: Test arm
Biological: Yellow Fever vaccine — STAMARIL, 1 dose (0.5 ml)
  Other Names: Stamaril

SUMMARY:
Epidemic viral diseases have become more prevalent in recent years. Among the various strategies to prevent such epidemics, vaccination is the most cost-effective. However, populations that are immunized are typically already exposed to multiple previous vaccinations or natural infections. Studies from this and other laboratories have revealed that pre-existing dengue antibodies can either inhibit or enhance subsequent dengue infection depending on the pre-existing antibody levels. While cross-reactive antibody is potentially pathogenic in dengue, how it impacts immune response to vaccination is unclear. Indeed, aggregated at the site of vaccination and the respective draining lymph nodes are antigen-presenting and immune regulatory cells that express Fc receptors and play pivotal roles in determining the magnitude and polarity of the immune response. Vaccine uptake by these antigen-presenting cells may thus be either inhibited or enhanced when vaccines are opsonized with cross-reactive antibodies.

In view of the limited knowledge on how cross-reactive antibodies affect vaccination outcome, investigators propose here a study that exploits the known cross reactivity between Japanese encephalitis (JE) virus antibody and yellow fever (YF) vaccine. Investigators hypothesize that cross-reactive antibodies impacts antibody response to YF at the point vaccination in a concentration-dependent manner by altering both vaccine uptake and the innate immune response by antigen presenting cells. Investigators will structure an open label clinical trial on sequential vaccination with JE and YF vaccines, with different time intervals between vaccinations. This would test immune response to YF vaccination in subjects with different titer of cross-reactive JE vaccine-derived antibodies.

DETAILED DESCRIPTION:
The primary objective of this clinical study is to examine the role of cross-reactive antibodies in modulating immune responses to vaccines.

1. Hypothesis: Antibody response to YF vaccination is influenced by the heterologous antibody titer at the point of YF vaccination.
2. Hypothesis : Heterologous antibody to YF affect magnitude of vaccine uptake through the Fc receptors and alters the quality and magnitude of the innate immune response following YF vaccination, which has been previously shown to predictive of immune response to YF vaccination.

Secondary objectives

1. To determine neutralizing antibody response to YF vaccination in human volunteers at different time intervals following a prior JE vaccination.
2. To characterize the innate immune response to YF vaccination at different time intervals after a prior JE vaccination.

A total of 100 healthy adults, pre-screened to be negative for anti-dengue antibodies will be enrolled upon written informed consent. 75 subjects in the test arm will received 2 doses of inactivated JE vaccine(Ixiaro), while 25 subjects in the control arm has no JE vaccination.

Subjects in the test arm will be sub-divided into 3 groups who receive YF17D:

Group1.YF vaccination 1-month post-JE vaccination Group 2.YF vaccination 4-months post-JE vaccination Group 3.YF vaccination 9-months post-JE vaccination Subjects in the control arm (group 4) will receive YF vaccination at the same time as group 1.

Blood sampling in relation to YF17D vaccination:

1. Pre-dose
2. 1-day after
3. 3-days after (+ 1 day)
4. 1-week after (± 2 days)
5. 1-month after (± 5 days)
6. 1-year after (± 14 days)

Primary end-point: Difference in geometric mean titre of YF17D neutralizing antibody.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female adults, 21-50 years of age at the time of screening.
* Negative for anti-dengue antibodies by ELISA.
* Subjects who are willing to comply with the requirements of the study protocol and scheduled visits. (e.g., completion of the subject diary, return for follow-up visits) and who are willing to make themselves available for the duration of the study, with access to a consistent means of telephone contact, which may be either at home or at the workplace, land line, or mobile, but NOT a pay phone or other multiple-user device (i.e. a common-use phone serving multiple rooms or apartments).
* Subjects who give written informed consent approved by the Ethical Review Board governing the site.
* Satisfactory baseline medical assessment as assessed by physical examination and a stable health status. The laboratory values must be within the normal range of the assessing site or show abnormalities that are deemed not clinically significant as judged by the investigator. A stable health status is defined as the absence of a health event satisfying the definition of a serious adverse event.
* Accessible vein the forearm for blood collection.
* Females of non-child bearing potential due to surgical sterilization (hysterectomy or bilateral oophorectomy or tubal ligation) or menopause.
* Female subjects of childbearing potential may be enrolled in the study

  1. if they have a negative urine pregnancy test on the day of screening and negative urine dipstick pregnancy tests at the days of the vaccinations
  2. if they use adequate, reliable contraception or abstain from sexual intercourse during the entire study for 1 year

Exclusion Criteria:

* Presence of acute infection in the preceding 7 days or presence of a temperature ≥ 38.0°C (oral temperature assessment), or acute symptoms greater than of "mild" severity on the scheduled date of first vaccination.
* History of severe drug and /or food allergies and/or known allergies to the trial product or its components.
* Any condition that, in the opinion of the investigator, would complicate or compromise the study or wellbeing of the subject.
* Woman who are pregnant or breast feeding.
* History or presence of cardiovascular, respiratory, hepatic, renal, gastrointestinal, neuropsychiatric, or immunosuppressive disorders that would be a risk factor when administered the IP.
* History of thymus gland disease.
* Diagnosed with cancer or on treatment for cancer within the 3 years prior to the screening.
* Evidence of clinically significant anaemia and other any significant active haematological disease, or having donated > 450 mL of blood within the past three months.
* Evidence of substance abuse, or previous substance abuse.
* Participation in a study involving administration of an investigational compound within the past four months, or planned participation during the duration of this study.
* Administration of any licensed vaccine, such as MMR and/or Chickenpox immunisation within 30 days before the first study vaccine dose.

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 84 (Actual)
Dates: Start 2013-10; Primary Completion 2015-06 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Difference in geometric mean neutralizing antibody titer to YF17D as measured by plaque reduction neutralization test (PRNT) in volunteers receiving YF vaccination with or without prior JE vaccination | 1-month and 1-year post YF17D vaccine

SECONDARY OUTCOMES:
Innate immune response to YF vaccination at different time intervals after a prior JE vaccination | transcriptional profiling of PBMC collected 1-day before, 1-, 3- and 7-days post YF17D vaccine

CONTACTS AND LOCATIONS:
Overall Officials: Jenny Low Guek Hong, Principal Investigator — Singapore General Hospital
Locations (1):
- Singhealth Investigational Medicine Unit, Singapore, Singapore

REFERENCES:
- [Derived] Low JG, Wijaya L, Li GK, Lim EY, Shum AK, Cheung YB, Ooi EE. The role of pre-existing cross-reactive antibodies in determining the efficacy of vaccination in humans: study protocol for a randomized controlled trial. Trials. 2015 Apr 10;16:147. doi: 10.1186/s13063-015-0651-z. PMID 25872531